CLINICAL TRIAL: NCT01017185
Title: Phase I Trial of Intratumoral Administration of HF10, A Replication Competent Herpes Simplex Virus Type 1, in Patients With Refractory Head and Neck Cancer or Solid Tumors With Cutaneous and/or Superficial Lesions
Brief Title: Study of HF10 in Patients With Refractory Head and Neck Cancer or Solid Tumors With Cutaneous and/or Superficial Lesions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takara Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M06-10083
Record Dates: First submitted 2009-11-18; First posted 2009-11-20 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2015-05

CONDITIONS: Refractory Head and Neck Cancer; Squamous Cell Carcinoma, Skin; Carcinoma of the Breast; Malignant Melanoma
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell; Breast Neoplasms; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oncolytic virotherapy, intratumoral injection of HF10 (Experimental)
  Interventions: Drug: HF10

INTERVENTIONS:
Drug: HF10

SUMMARY:
The purpose of this study is to determine whether HF10 is safe and effective in the treatment of head and neck cancer or solid tumors with cutaneous and/or superficial lesions.

DETAILED DESCRIPTION:
This is an open label, non-randomized, multicenter, two-stage, dose escalation Phase I study evaluating single and repeated intratumoral injections of the oncolytic virus, HF10, in patients with refractory head and neck cancer, or solid tumors with cutaneous and/or superficial lesions (e.g., squamous cell carcinoma of the skin, carcinoma of the breast, and malignant melanoma).

Stage 1: Stage 1 of the study will investigate dose escalation of a single intratumoral injection over the following dose levels: 1 x 10^5 TCID50, 3 x 10^5 TCID50, 1 x 10^6 TCID50, and 1 x 10^7 TCID50. In Stage 1, it is planned that 3 patients will be enrolled per single dose cohort. Within each single dose cohort, accrual will temporarily be suspended after the first patient is entered and the patient will be followed for safety and for viral distribution and elimination. The patients in Stage 1 must be seropositive for HSV-1.

Stage 2: Stage 2 will evaluate repeated intratumoral injections of HF10 at dose levels of 1 x 10^6 TCID50/dose and 1 x 10^7 TCID50/dose. Three patients will be enrolled in each of the repeated dose cohorts. In Stage 2, the first patient treated in each repeated dose cohort must be seropositive for HSV-1. Patients in the repeated dose cohort will receive a total of four intratumoral injections in the same lesion.

Following completion of dosing in the repeated dose cohorts, an expansion cohort of three additional patients will be treated at the highest tolerated dose level.

ELIGIBILITY:
Inclusion Criteria

* Patients must have histologically confirmed solid tumors that have failed standard therapies (surgery, chemotherapy, radiotherapy, or endocrine therapy) and for which no curative options exist, including, but not limited to:

  * Squamous cell carcinoma of the head and neck
  * Squamous cell carcinoma of the skin
  * Carcinoma of the breast
  * Malignant melanoma
* Patients may have had any kind and number of prior cancer therapies.
* Patients must have measurable non-visceral lesions that are evaluable by the RECIST method
* The tumor mass to be treated must be non-visceral and adequate for injection (i.e., more than 2 cm away from major vascular structures) and measurement by RECIST.
* Patients in Stage 1 must be seropositive for HSV-1.
* The first patient enrolled into each cohort in Stage 2 must be seropositive for HSV-1.
* Patients must be ≥ 18 years of age.
* Patients must have a life expectancy ≥ 12 weeks
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Patients must have adequate hepatic function, as defined as

  * Total bilirubin levels ≤ 1.5 x upper limit of normal (ULN)
  * AST/ALT levels ≤ 2.5 x ULN, or ≤ 5 x ULN if liver metastases are present
* Patients must have adequate renal function as defined as serum creatinine ≤ 1.5 x ULN or creatinine clearance (calculated) ≥ 60 mL/min/1.73 m2 for patients with creatinine > 1.5 x ULN
* Patients must have adequate bone marrow function, as defined as

  * Absolute neutrophil count ≥ 1,500/μL and
  * Platelet count ≥ 100,000/μL
* Patients must have no known bleeding diathesis or coagulopathy that would make intratumoral injection or biopsy unsafe.
* Men and women of childbearing potential must agree to use adequate contraception prior to study entry and for up to six months.
* Females of childbearing potential must have a negative urine or serum pregnancy test within one week prior to start of treatment.
* Patients must be able to understand and willing to sign a written informed consent document.

Exclusion Criteria

* Patients receiving chemotherapy or radiotherapy within 4 weeks of injection of HF10, or adverse events > Grade 1, except alopecia, resulting from agents administered more than 4 weeks prior to HF10 injection.
* Patients with a history of significant tumor bleeding, or coagulation or bleeding disorders.
* Patients with nasopharyngeal tumors.
* Patients with deep (below the platysma muscle layer) ulcerative tumors.
* Patients with target tumors that could potentially invade a major vascular structure(s) (e.g., innominate artery, carotid artery), based on unequivocal imaging findings, as determined by a radiologist.
* Patients with Grade ≥ 1 pre-existing neurologic abnormalities (CTCAE version 3.0).
* Patients who have been hospitalized for emergent conditions requiring inpatient evaluation, treatment or procedure during the 30 days prior to entry on study. In addition, emergent conditions requiring inpatient evaluation, treatment or procedure must have resolved or be medically stable and not severe for 30 days prior to entry on study.
* Patients with clinically evident Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), Hepatitis C virus (HCV), or Epstein-Barr virus (EBV) infection. Patients will be tested for HIV during pre-treatment screening.
* Patients receiving steroids or immunosuppressive agents, e.g., for rheumatoid arthritis
* Concurrent use of any other investigational agents.
* Presence or history of central nervous system metastasis.
* Pregnant or breastfeeding women;women desiring to become pregnant within the timeframe of the study are also excluded.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-08; Primary Completion 2014-05 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Assessment of the local tumor response of the HF10-injected tumor by a modified target Response Evaluation Criteria In Solid Tumors (RECIST) method | one year

SECONDARY OUTCOMES:
Adverse events, vital signs, electrocardiogram(ECG), clinical laboratory tests, and physical exercise | one year
Histological tumor response by biopsy | one year
Overall tumor response of the HF10-injected tumor plus additional non-injected target tumors. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Ferris, MD, PhD, Principal Investigator — Division of Head and Neck Cancer Surgery, University of Pittsburgh Cancer Institute
Locations (5):
- United States (5):
  - Montefiore Medical Center, The Bronx, New York
  - Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah